CLINICAL TRIAL: NCT00472693
Title: A Phase II Trial of Bevacizumab and ABI-007 (Abraxane) as Second-line Therapy in Her-2 Negative, Hormone Receptor Negative Metastatic Breast Cancer
Brief Title: Bevacizumab and Abraxane as Second-line Therapy in Triple Negative Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 02106
Record Dates: First submitted 2007-05-11; First posted 2007-05-14 (Estimated); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Metastatic breast cancer; Second-Line Therapy; Triple Negative; Her-2 negative; Hormone receptor negative; Abraxane; Bevacizumab
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bevacizumab and ABI-007 (Abraxane) (Experimental): Bevacizumab and ABI-007 (Abraxane)
  Interventions: Drug: Bevacizumab, Abraxane

INTERVENTIONS:
Drug: Bevacizumab, Abraxane — Bevacizumab, 10 mg/m2 IV days 1 and 15; ABI-007, 100 mg/m2 IV days 1, 8, 15 of each 28 day cycle. Continue treatment until disease progression, patient withdrawal or unacceptable toxicities.

SUMMARY:
The purpose of this study is to determine whether the addition of bevacizumab to Abraxane as second-line therapy in Her-2 negative, hormone receptor negative metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 18 years or older and able to give informed consent.
* Histologically- or cytologically-proven adenocarcinoma of the breast at time of first diagnosis
* ECOG performance status 0 or 1
* Life expectancy > 12 weeks
* Stage IV disease and have at least one lesion measurable by standard RECIST criteria
* Disease progression after at least one prior chemotherapy regimen for metastatic disease or within 12 months of adjuvant chemotherapy initiation.
* All chemotherapy must be stopped > 2 weeks before enrollment.
* Primary or metastatic tumor must be negative for estrogen and progesterone receptor expression. Testing must be done in a CLIA-approved laboratory.
* Primary or metastatic tumor must have 0 or 1+ staining for HER2/neu identified immunohistochemically (IHC), by an approved method using one of the standard monoclonal or polyclonal antibodies (HercepTest, cb-11, PAb1, or TAB250), or if FISH status is known, it must be negative. Testing must be done in a CLIA-approved laboratory.
* Left ventricular ejection fraction must be >= institutional lower limit of normal as determined by MUGA or echocardiogram
* Patient must be able to comply with treatment and follow-up procedures:
* Adequate bone marrow, liver and renal function; Absolute neutrophil count >= 1500/mm3; Hemoglobin >= 10 g/dl; Platelet count >= 100,000/mm3; Creatinine <= 2.0; PTT and either INR or PT < 1.5x normal; Total bilirubin <= 1.5 X upper limit of normal; AST, ALT, and alkaline phosphatase <= 2 X upper limit of normal (or <= 5X upper limit of normal if known liver metastases)
* If female is of childbearing potential, pregnancy test must be negative and patient must be willing to use effective contraception while on treatment and for at least 3 months after the last dose of study medication

Exclusion Criteria:

* Prior treatment with VEGF targeted therapy
* Prior taxane therapy for metastatic disease or for adjuvant therapy within the previous 12 months
* History of prior cancer, excluding carcinoma in situ of the cervix and non-melanoma skin cancers
* Known CNS disease
* Inadequately controlled hypertension (defined as systolic blood pressure>150 and/or diastolic blood pressure>100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure
* History of myocardial infarction or unstable angina within 6 months prior to study enrollment
* History of stroke or transient ischemic attack within 6 months prior to study enrollment
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study enrollment or anticipation of need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to study enrollment
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to study enrollment
* Serious, non-healing wound, ulcer or bone fracture
* Proteinuria at screening as demonstrated by either: Urine protein:creatinine (UPC) ratio >1.0 at screening OR Urine dipstick for proteinuria >2+ (patients discovered to have >2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate <1g of protein in 24 hours to be eligible)
* Patients with active infection
* Women who are pregnant or lactating
* Radiation therapy within 3 weeks of study entry
* Patients with hypersensitivity to ABI-007, Chinese hamster ovary cell products, or other recombinant human antibodies
* Baseline neuropathy > grade 2
* Participation in an investigational study of an antineoplastic agent within 4 weeks of first infusion of this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To determine progression-free survival among women receiving bevacizumab + ABI-007 given as second-line combination therapy for hormone receptive negative, Her-2 negative metastatic breast cancer. | Study Completion

SECONDARY OUTCOMES:
To determine the overall response rate to bevacizumab + ABI-007 in this study population. | Study completion
To determine the toxicity of bevacizumab + ABI-007 in this study population. | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, M.D., Principal Investigator — Abramson Cancer Center of University of Pennsylvania
Locations (1):
- Abramson Cancer Center at University of Pennsylvania, Philadelphia, Pennsylvania, United States